CLINICAL TRIAL: NCT02682368
Title: Multicentric Point of Care UltraSound by Surgeons Trial
Acronym: POCUSS
Status: Completed | Type: Observational
Sponsor: Connolly Hospital Blanchardstown (Other)
Collaborators: Royal College of Surgeons, Ireland (Other); Modular UltraSound ESTES Course (MUSEC) (Unknown); European Society for Trauma and Emergency Surgery (Other)
Responsible Party: Principal Investigator, Daniel B Dumbrava, MD, General Surgery Trainee, Connolly Hospital Blanchardstown
Other Study IDs: 15190484; 255774 (Other: Trademark act 1996, Irish Patent Office)
Record Dates: First submitted 2016-01-25; First posted 2016-02-15 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Biliary Disease; Gallstone; Cholecystitis, Acute; Diverticulitis, Colonic; Abscess Pelvic
Keywords: Surgeon performed ultrasound; Point of care ultrasound
MeSH Terms: conditions — Gallbladder Diseases; Gallstones; Cholecystitis; Diverticulitis, Colonic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- POCUSS Trial-1 Acute Biliary Disease: Patients with suspected biliary pathology which will undergo POCUS. The results will be compared to the subsequent findings by imagistic means or at time of surgery.
  Interventions: Diagnostic Test: Point of Care Ultrasound by Surgeons (POCUSS)
- POCUSS Trial-2 Acute Diverticulitis: Patients with suspected diverticulitis will undergo POCUS. The results will be compared to the subsequent findings by imagistic means or at time of surgery.
  Interventions: Diagnostic Test: Point of Care Ultrasound by Surgeons (POCUSS)
- Radiology Report: Departmental imaging and reports.
  Interventions: Diagnostic Test: Radiology report
- Surgical diagnostic: Intraoperative findings of patients that undergo emergency surgery.
  Interventions: Procedure: Surgery-Intra-operative findings

INTERVENTIONS:
Diagnostic Test: Point of Care Ultrasound by Surgeons (POCUSS) — POCUSS-1. To identify the gallbladder and it's contents, complications and perform measurements, elicit sonographic Murphy.
  POCUSS-2: To perform focused left lower quadrant sonography and identify bowel wall thickness, diverticulae, measure the colonic wall thickness, assess pericolic fat and detect possible complications; evaluate sensibility on graded compression.
  Other Names: Sonos®, BK Ultrasound®
  Groups: POCUSS Trial-1 Acute Biliary Disease; POCUSS Trial-2 Acute Diverticulitis
Diagnostic Test: Radiology report — Radiologist report compared to the point of care ultrasound impression.
  Other Names: NIMIS: The National Integrated Medical Imaging System
  Groups: Radiology Report
Procedure: Surgery-Intra-operative findings — Intra-operative findings compared to the previously performed point of care ultrasound.
  Groups: Surgical diagnostic

SUMMARY:
Acute gallbladder pathology and acute diverticulitis are common conditions met in emergency departments and comprise the bulk of admissions throughout general surgical calls. Both entities need imagistic description to tailor further management, which may be not readily available at the moment of patient's presentation. These delays may lose the window of opportunity for timed, quality decision making and may induce increased length of stay and subsequent increased costs.

Ultrasound scanning has become very popular over the last half century and the equipment has become more compact, of a higher quality and less expensive, which has facilitated the growth of point-of-care ultrasonography - POCUS - that is, ultrasound performed and interpreted by the clinician at the bedside. The concept of an 'ultrasound stethoscope' is rapidly moving from theory to reality.

There are a number of studies and case reports that are highlighting the advantages of POCUS, but still common grounds need to be sought after. Some countries, like USA and Germany, incorporate basic ultrasound in their resident's curriculum among different specialties.

In the author's knowledge and based on the literature, there are a few-second-to-none studies regarding POCUS involving strictly the surgeons. The hypothesis of this study is that, surgeon performed ultrasound can be as accurate as the radiologists' findings for basic diagnostics in the aforementioned pathology, leading to real time decision making in the benefit of the patient.

The closing remark is that by learning and doing these procedures the surgeon performing POCUS doesn't undermine his/her radiologist colleague's authority and skill. The big picture is that some basic tasks are transferrable and if used in an appropriate and methodical manner the final common goal - the benefit of the patient - is readily achieved.

DETAILED DESCRIPTION:
The study was accepted as a Master of Surgery Thesis by Research (MCh) at the Royal College of Surgeons in Ireland (RCSI)

There will be two parallel studies done at the same time:

1. POCUSS-1 for acute biliary disease
2. POCUSS-2 for suspected diverticulitis

STUDY DESIGN

1. Patients with suspected acute biliary disease or acute diverticulitis will undergo POCUS performed by the surgeons enrolled in the study.

   These patients are recruited from either
   1. emergency department
   2. outpatients clinic
   3. ward consults
2. Patients will have the procedure explained to them and then will receive a leaflet with the same information will be handed over. Consent will be obtained (verbal and written) from the patients that wish to be enrolled in the study.
3. POCUS is performed and data recorded on REDCap®.

4a. The same patients will have a departmental imagistic investigation (ultrasound, CT) reported by qualified radiologists.

4b. In the event of emergency surgery without prior departmental imaging, POCUS will be compared to the intra-operative findings.

5. Data will be collected and stored anonymously and processed with REDCap, Microsoft Excel, IMB SPSS, R-studio

DISCLAIMER:

Specific for this study, patient data will be anonymous and in line with General Data Protection Regulation (GDPR) (EU) 2016/679 law. Data protection is designed by default. There will be NO patients' personal name, surname, home address or date of birth needed or uploaded. Each patient will be represented by an unique identification number provided by the hospital. Only gender and age will be recorded as these will be necessary for the final data analysis and results. Once the study has finished, the data will be erased.

The same rules will be applied in hospitals from other countries that will get involved in the study.

ELIGIBILITY:
POCUS-1 Inclusion Criteria - adapted after Tokyo Guidelines 2018

1. RUQ mass/pain/tenderness
2. Murphy's Sign
3. Fever
4. Elevated WBC
5. Elevated CRP
6. Deranged liver function tests
7. Jaundice

POCUS-2 Inclusion Criteria

1. Left iliac fossa tenderness and/or palpable mass
2. Fever
3. Elevated WBC
4. Elevated CRP
5. Peritonism - Left lower quadrant / hypogastrium
6. Per rectum bleeding/mucus discharge

POCUSS-1 and 2 Exclusion Criteria:

1. Age under 18 (ethical and consent issues)
2. Pregnancy
3. Obesity (BMI ≥ 30)-difficulty in performing USS
4. Previously documented gallstones within the last 2 months for non-critical presentations
5. Previously documented diverticulitis within the last 2 months for non-critical presentations
6. POCUS performed after official report (for training purposes)
7. Previous colonic resection, particularly left sided or sigmoid colon.
8. Previous cholecystectomy

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Emergency Department with a clinical suspicion of acute cholecystitis and/or acute sigmoid diverticulitis.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity POCUS | Up to 3 years, after the all the patients are included
  Sensitivity was defined as the number of patients with a positive detection at POCUS of acute biliary disease or acute diverticulitis divided by the number of patients with pathological findings of the gallbladder or bowel as a final diagnosis.
Specificity POCUS | Up to 3 years, after the all the patients are included
  Specificity was defined as the number of patients with a negative POCUS for cholecystitis or diverticulitis, divided by the number of patients without pathological findings.
Positive predictive value | Up to 3 years, after the all the patients are included
  The number of patients with a true-positive detection at POCUS of gallbladder or bowel alteration divided by the total number of patients with a positive detection at POCUS.
Negative predictive value | Up to 3 years, after the all the patients are included
  The number of patients with a true-negative detection at POCUS of gallbladder or bowel alteration divided by the total number of patients with a negative detection at ultrasound.
POCUS and radiology/surgery correlation | Up to 3 years, after the all the patients are included
  Cohen's Kappa for agreement between POCUS and radiology

SECONDARY OUTCOMES:
Radiology turnaround time | Up to 1 week
  Time difference (in hours) between radiologist report and POCUS. For each participant date and time will be recorded in REDCap for both POCUS and radiology report. Simple arithmetic subtraction will be used as an equation cell (datediff). Then mean and median will be calculated to include all patients in the study.
Surgery turnaround time | Between 6 and 48 hours, when emergency surgery would be expected
  Time difference (in hours) between the start of surgery and POCUS. For each participant date and time will be recorded in REDCap for both POCUS and surgical intervention. Simple arithmetic subtraction will be used in a calculation cell (datediff). Then mean and median will be calculated to include all patients in the study.
Likelihood ratio | Up to 3 years
  Likelihood ratio for a positive test result = sensitivity/(1 - specificity)
  Likelihood ratio for a negative test result = (1 - sensitivity)/specificity

CONTACTS AND LOCATIONS:
Overall Officials: Thomas N Walsh, MCh MD FRCSI, Study Director — Connolly Hospital Blanchardstown; Royal College of Surgeons in Ireland; Gary A Bass, MBBCh MSc MRCS, Study Chair — Connolly Hospital Blanchardstown; Royal College of Surgeons in Ireland; Daniel B Dumbrava, MBBCh, Principal Investigator — Connolly Hospital Blanchardstown; Royal College of Surgeons in Ireland
Locations (5):
- Connolly Hospital Blanchardstown, Dublin, Dublin 15, Ireland
- Italy (2):
  - General Surgery Dept, Minimally Invasive Surgery Unit, Policlinico San Pietro, Ponte San Pietro, Bergamo
  - General Surgery Department, ASUITS, Cattinara Hospital, Trieste
- Centro Hospitalar Tondela Viseu - Serviço de Cirurgia Geral - Unidade de Cirurgia HBP, Viseu, Centro Region, Portugal
- Torrevieja University Hospital, Torrevieja, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No
Specific for this study, patient data will be anonymous and in line with General Data Protection Regulation (GDPR) (EU) 2016/679 law. Data protection is designed by default. There will be NO patients' personal name, surname, home address or date of birth needed or uploaded. Once the study has finished, the working data will be erased. Only the processed data and statistical analysis will be preserved.

REFERENCES:
- [Derived] Dumbrava BD, Bass GA, Jumean A, Birido N, Corbally M, Pereira J, Biloslavo A, Zago M, Walsh TN. The Accuracy of Point-of-Care Ultrasound (POCUS) in Acute Gallbladder Disease. Diagnostics (Basel). 2023 Mar 26;13(7):1248. doi: 10.3390/diagnostics13071248. PMID 37046466
- [Derived] Dumbrava BD, Abdulla HS, Pereira J, Biloslavo A, Zago M, Hashem JH, Kumar N, Corbally M, Bass GA, Walsh TN. Surgeon-Performed Point-of-Care Ultrasound in the Diagnosis of Acute Sigmoid Diverticulitis: A Pragmatic Prospective Multicenter Cohort Study. Cureus. 2023 Jan 3;15(1):e33292. doi: 10.7759/cureus.33292. eCollection 2023 Jan. PMID 36741667